CLINICAL TRIAL: NCT05766215
Title: Influence of Nurse-led Therapeutic Patient Education on Glycemic Control and Knowledge of Patients With Type 1 Diabetes Mellitus in Hospital Transition: a Quasi-experimental Trial
Brief Title: Nurse-led Therapeutic Education Effects in Glycemic Control and Knowledge of Type 1 Diabetes Mellitus Patients Under Hospital Transition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Pilar Santa Cruz Álvarez, Enfermera de Práctica Avanzada (EPA), Hospitales Universitarios Virgen del Rocío
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MPSA-ETDT-2022
Record Dates: First submitted 2022-12-22; First posted 2023-03-13 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Nurse's Role
Keywords: type 1 diabetes mellitus; health education; glycated hemoglobin A; health-related knowledge
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic patients education (Experimental): 3 sessions of structured therapeutic patient education (TPE) in which diet, exercise, alcohol abuse and insulin or pharmacological treatment management advise is given.
  Interventions: Behavioral: Therapeutic Education

INTERVENTIONS:
Behavioral: Therapeutic Education — It consists of four structured phases: 1. Welcome nurse visit, 2. Diabetologic education course adapted to the detected needs, 3. Individualized follow-up through alternating quarterly appointments between nurses and endocrine physician, 4. Evaluation and discharge of the program

SUMMARY:
The goal of this interventional quasiexperimental study is to learn about the influence of therapeutic education carried out by nurses in the management and knowledge of patients with T1DM. Participants will be:

Given several therapeutic education sessions. Evaluated using different questionnaires and anthropometric measures.

DETAILED DESCRIPTION:
The main objective of the study will be to determine the influence of therapeutic education carried out by nurses in the management and knowledge of patients with T1DM who will make a hospital transition. The research design will be a single-blind, nonrandomized, quasi-experimental, single-center, 1-group controlled study .

It will be developed at the Center for Diagnosis and Treatment (CDT) of the Virgen del Rocío University Hospital (HUVR), in Seville (Spain). The participant selection process will be carried out considering that only 13 adolescents 17 and 18 years and younger with T1DM, belonging to the reference hospital area, will transit from the Children's Hospital to the Adult Hospital. It is estimated that the study will have a sample of a minimum of n=10, which will be studied over 12 months.

Given the existing bibliography about the benefits of this intervention , 1 it is expected that the glycosylated hemoglobin (HbA1c) of patients will be less than 7%, which together with the Self-Management Adherence Questionnaire for Diabetes Treatment (SCI-R. es) 2 represents that patients perform adequate management of their disease. The Survey of Eating Problems in Diabetes Summary Questionnaire (EPAD-R) 3 will be used to assess their eating behavior. An improvement in people's knowledge regarding hypoglycemia is also sought, measured with the Clarke test 4 ; and an improvement in the quality of life, measured with the SF-12 questionnaire 5 and family support with the Apgar test 6 .

The therapeutic plan consists of preparing the process prior to discharge from the pediatric center, transferring to the adult hospital with a clinical and educational report and a previously arranged visit to the new unit. The heads of both teams coordinate the structure and the transition process with regular meetings. From the Adult Diabetes Day Hospital, a joint visit is reserved with the endocrinologist and the nurse educator. They are integrated into a 12-month therapeutic care and education program. It consists of four structured phases: 1. Welcome nurse visit, 2. Diabetologic education course adapted to the detected needs, 3. Individualized follow-up through alternating quarterly appointments between nurses and endocrine physician, 4. Evaluation and discharge of the program.

At the beginning (baseline visit), at 3 and 12 months the following variables are recorded:

1. Age (years), sex (female/male), T1DM evolution (years).
2. Treatment type (basal-bolus/insulin pump). Sensor usage time (>80%)
3. Metabolic control: HbA1C (mg/ dL ), Time in Range (TIR), Time Above Range (TAR), Time Below Range (TBR), Coefficient of Variation (CV), Mean Glucose (GMI), weight (Kg), height (cm), BMI (Kg/m 2 ).
4. Perception of quality of life. Test SF-12, of 12 questions.
5. Perception of symptoms of hypoglycemia. Clarke test, 8 questions.
6. Eating behavior, with the EPAD-R test, of 16 questions.
7. Adherence to diabetes treatment. SCI-R.es test. The results analysis plan will be carried out using Microsoft Excel, SPSS or R Commander computer programs , in which the relationships between the descriptive statistics extracted from the screened data will be explored to prevent duplicates. The same digital tools will be used to guarantee the protection of the data and variables collected. This aspect is detailed in the attached informed consent.

Regarding the ethical and legal aspects of the study, it is worth mentioning the benefit in disease management, quality of life and general satisfaction that the protocolized follow-up will cause in adolescents. No risk to the psychosocial integrity of the population involved in the study has been detected.

The necessary facilities will be the Education Classroom of the HUVR Diabetes Day Hospital, computer support through 2 computers, paper resources for the questionnaires, 2 nurses and 1 endocrinologist will be necessary as human resources. The authors declare the absence of funding or conflict of interest for the development of the research.

ELIGIBILITY:
Inclusion Criteria:

* Age 17 years.

Exclusion Criteria:

* Unable to give informed consent.

Ages: 17 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 13 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2024-01-22 (Estimated); Study Completion 2024-12-22 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin. | 12 months
  HbA1c
Time in Range | 12 months
  TIR
Time above range | 12 months
  TAR
Time below range | 12 months
  TBR
Coefficient of variation | 12 months
  CV
Glucose Management Indicator | 12 months
  GMI
Weight | 12 months
  Kg
Height | 12 months
  cm
Body Mass Index | 12 months
  BMI

SECONDARY OUTCOMES:
Perception of quality of life. | 12 months
  SF-12
Perception of symptoms of hypoglycemia | 12 months
  Clarke
Eating behavior, | 12 months
  EPAD-R
Adherence to diabetes treatment | 12 months
  SCI-R

OTHER OUTCOMES:
Treatment type | 12 months
  basal-bonus, insulin pump, sensor usage range
Demographical information | 12 months
  Age (years), sex (female/male), T1DM evolution (years).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospitales Universitarios Virgen del Rocío, Seville, Spain

IPD SHARING:
Plan to Share IPD: No